CLINICAL TRIAL: NCT02406885
Title: APB Study: Apixaban Pharmacokinetics in Bariatric Patients
Brief Title: Apixaban Pharmacokinetics in Bariatric Patients (APB)
Acronym: APB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00035495
Record Dates: First submitted 2015-02-05; First posted 2015-04-02 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Bariatric Surgery; Obesity
MeSH Terms: conditions — Obesity | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APB study: Apixaban Pharmacokinetics in VSG (Active Comparator): To determine the durability or change in pharmacokinetics and pharmacodynamics of apixaban in patients with a body mass index (BMI) of 35 kg/m2 or greater pre vs. post surgery for patients undergoing vertical sleeve gastrectomy
  Interventions: Drug: Apixaban
- APB study: Apixaban Pharmacokinetics in RYGB (Active Comparator): To determine the durability or change in pharmacokinetics and pharmacodynamics of apixaban in patients with a body mass index (BMI) of 35 kg/m2 or greater pre vs. post surgery for patients undergoing Roux-en Y gastric bypass.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — New Oral Anticoagulants (NOACs) are currently available for prophylaxis against venous thromboembolism in patients undergoing total hip or knee replacement surgery.
  Other Names: Eliquis

SUMMARY:
The Center for Bariatric Surgery is interested in conducting a pharmacokinetic study of apixaban (an oral anticoagulant with FDA approval for use of venous thrombo embolism (VTE) prophylaxis and treatment) in the obese adult population to determine if bariatric surgery influences apixaban exposure. More interesting would be to see how the dose may need to change pre- vs. post-bariatric surgery (this will be important for physicians as more and more patients undergo this procedure worldwide and many may require anticoagulation in their future healthcare).

Physicians and surgeons are very interested in oral anticoagulants for this special patient population. To date, there is no approved dosing for the obese patient (especially when considering surgical intervention such as bariatric surgery).

Primary outcome variable.

To determine the durability or change in pharmacokinetics and pharmacodynamics of apixaban in patients with a body mass index (BMI) of 35 kg/m2 or greater following one of two bariatric surgical procedures (pre-operative versus post-operative vertical sleeve gastrectomy or Roux-en-Y gastric bypass patients).

Secondary outcome variables.

1. To compare/contrast the pharmacokinetics and pharmacodynamics of apixaban in bariatric surgical patients who have undergone RYGB vs. VSG.
2. To determine how the pharmacokinetics of the drug may differ when there is significant post-operative surgical weight loss (>40% estimated excess body weight) 12 to 18 months following surgery versus those patients who have suboptimal weight loss following bariatric surgery (< 40% of estimated excess body weight).

DETAILED DESCRIPTION:
Obesity is now the leading health problem of the 21st century. Weight reduction by conservative methods including diet and exercise has had poor success rates. There has been a substantial increase in the use of bariatric surgery to provide sustained weight loss and thus a reduction in the medical comorbidities that are associated with obesity. However, because these procedures may alter the anatomical and physiological aspects of the gastrointestinal system, there is a possibility of altered pharmacokinetics to medications particularly when taken orally. Furthermore, patients typically lose anywhere from 50 to 75% of their estimated excess body mass approximately one to two years following surgery. This successful therapeutic outcome of the surgery may be causing long term changes in the pharmacokinetics that are independent of any direct anatomical or physiologic changes induced by the procedure.

Physicians and surgeons are very interested in oral anticoagulants for this special patient population. To date, there is no approved dosing for the obese patient (especially when considering surgical intervention such as bariatric surgery). VTE is one of the top two causes of morbidity and mortality in the bariatric surgical patient. In the ninth edition of the Antithrombotic Therapy and Prevention of Thrombosis guideline published by the American College of Chest Physicians (1), it is reported that virtually all bariatric surgical patients have at least a moderate risk of VTE, with many patients at high risk. (2) The approach to VTE prophylaxis used by most bariatric surgeons today is a combination of non-invasive and pharmacologic techniques, including sequential compression devices, anti-embolic stockings, anticoagulation, and early ambulation. Traditionally VTE prophylaxis has been accomplished with subcutaneous injection however with the introduction of new oral anticoagulant medications many practitioners are using these anticoagulants without demonstration of effectiveness in this population.

The Johns Hopkins Center for Bariatric Surgery is interested in conducting a pharmacokinetic study of apixaban (an oral anticoagulant with FDA approval for use of VTE prophylaxis and treatment) in the obese adult population to determine if bariatric surgery influences apixaban exposure. More interesting would be to see how the dose may need to change pre- vs. post-bariatric surgery (this will be important for physicians as more and more patients undergo this procedure worldwide and many may require anticoagulation in their future healthcare).

Specific Aim 1: To determine the pharmacokinetics of apixaban in obese patients scheduled to have bariatric surgery with a body mass index (BMI) of 35 kg/m2 or greater.

Hypothesis 1a: Obese patients prior to bariatric surgical intervention, compared to normal weight historical controls, will have a decrease in both Cmax and area under the curve (AUC) when given a single dose of 5 mg of apixaban.

Specific Aim 2: To determine the pharmacokinetics of apixaban in the bariatric surgical patient who has undergone Roux-en Y gastric bypass (RYGB) or Vertical Sleeve Gastrectomy (VSG) at 1, 6, 12 and 18 months post-op.

Hypothesis 2a: Patients who have recently undergone RYGB surgery (1 month post-op) will have a decrease in both the Cmax and AUC, relative to pre-op values, when given a single dose of 5 mg of apixaban.

Hypothesis 2b: Patients who have recently undergone VSG surgery (1 month post-op) will have a decrease in both the Cmax and AUC, relative to pre-op values, when given a single dose of 5 mg of apixaban. The magnitude of the decrease in Cmax and AUC will be less than that seen in RYGB patients.

Rationale: Anatomic alteration of the GI tract will immediately reduce absorption in all post-operative bariatric patients. In RYGB patients, the attenuated small bowel and altered bile acid composition will lead to decreased absorption of the drug, whereas in sleeve gastrectomy patients prolonged gastric emptying may affect pharmacokinetics.

These findings will be important when considering the use of apixaban as an oral anticoagulation option for perioperative VTE prophylaxis in the bariatric population, both in the acute hospital setting and after discharge in patients requiring extended VTE prophylaxis or treatment.

Hypothesis 2c: After undergoing bariatric surgery, patients at 6, 12, and 18 months post-op will have an increase in Cmax and AUC, relative to pre-op values, when given a single dose of 5 mg of apixaban.

Hypothesis 2d: After undergoing RYGB, patients at 6, 12, and 18 months post-op will have a greater increase in both Cmax and AUC, relative to pre-op values, than VSG patients relative to pre-op values when given a single dose of 5 mg of apixaban.

Rationale: Patients who are 6 to 18 months post-bariatric surgery generally have a 30-40% decrease in excess body weight. This decrease in body weight reduces volume of distribution of drug, potentially affecting Cmax. Results of the published Phase 1 apixaban study found that exposure to a dose of apixaban was inversely related to body weight. Therefore, the investigators should expect higher plasma levels of apixaban in patients who are 6 to 18 months post-bariatric surgery when compared to pre-op values.

Findings of the Phase I study (3,4) An open-label, parallel-group, non-randomized, single-dose study in healthy male and female subjects was conducted to assess the effects of body weight on the pharmacokinetics of a single 10 mg dose of apixaban. Following screening, patients were enrolled in one of three groups: low body weight (≤50kg, N=18), normal body weight (65-85kg, N=18) or high body weight (≥120kg, N=19).

Compared to normal body weight:

* There was a 27% increase in Cmax and 20% increase in AUC in patients with low body weight
* There was a 31% decrease in Cmax and 23% decrease in AUC in patients with high body weight

The effect of RYGB vs. sleeve gastrectomy on long-term pharmacokinetics is difficult to predict because of the opposing effects of greater weight loss with reduced absorption in the RYGB patient.

These findings will be important when considering apixaban as an oral medication for long-term post-op bariatric patients who may require anticoagulation for stroke, myocardial infarction, atrial fibrillation or orthopedic procedures such as hip or knee replacements. (5, 6)

Specific Aim 3: To measure the effect of apixaban on Factor Xa activity (chromogenic anti-Xa activity assay) in bariatric surgical patients pre-operatively then at 1, 6, 12 and 18 months post-operatively.

Hypothesis 3a: In spite of the changes in pharmacokinetics, the pharmacodynamics response (measured with a chromogenic anti-Xa activity assay) will not differ by more than 10% in comparing pre-surgical response to that at 1, 6, 12 and 18 months after surgery.

Rationale: The changes in pharmacokinetics should not lead to a different concentration-response relationship in the chromogenic anti- Xa activity of individual patients following dosing with apixaban 5 mg. Were there to be a significant change in pharmacodynamics, other factors due to the altered anatomy or substantial weight loss would need to be invoked to explain that altered relationship.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 65 years old with a BMI of 35 kg/m2 or greater who will be undergoing bariatric surgery (VSG and RYGB)
* Signed written informed consent
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
* Women must not be breastfeeding

Exclusion Criteria:

* History of documented clotting/coagulation disorder
* History of cancer (within the last year)
* Any diagnosis requiring anti-coagulation
* History of hypersensitivity reaction to apixaban
* Active clinically significant bleeding
* Creatinine > 1.5 mg/dL
* Participants currently receiving any type of anticoagulation or blood thinning medications, including heparin, low molecular weight heparins, Plavix, aspirin, NSAIDS
* Participant who is taking any of the excluded medications

  * Combined P-glycoprotein and strong cytochrome P450 (CYP) 3A4 inhibitor
  * Combined P-glycoprotein and moderate CYP 3A4 inhibitor
  * Combined P-glycoprotein inducer and strong CYP 3A4 inducer
  * Inducers of p-glycoprotein
  * Strong inducers of CYP 3A4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Petty, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Center for Bariatric Surgery, Baltimore, Maryland, United States

REFERENCES:
- [Background] Frost C, Wang J, Nepal S, Schuster A, Barrett YC, Mosqueda-Garcia R, Reeves RA, LaCreta F. Apixaban, an oral, direct factor Xa inhibitor: single dose safety, pharmacokinetics, pharmacodynamics and food effect in healthy subjects. Br J Clin Pharmacol. 2013 Feb;75(2):476-87. doi: 10.1111/j.1365-2125.2012.04369.x. PMID 22759198

RESULTS

PARTICIPANT FLOW:
Groups:
- APB Study: Apixaban Pharmacokinetics in RYGB: To determine the durability or change in pharmacokinetics and pharmacodynamics of apixaban in patients with a body mass index (BMI) of 35 kg/m2 or greater pre vs. post surgery for patients undergoing Roux-en Y gastric bypass (RYGB).
  Apixaban: New Oral Anticoagulants (NOACs) are currently available for prophylaxis against venous thromboembolism in patients undergoing total hip or knee replacement surgery.
- APB Study: Apixaban Pharmacokinetics in VSG: To determine the durability or change in pharmacokinetics and pharmacodynamics of apixaban in patients with a body mass index (BMI) of 35 kg/m2 or greater pre vs. post surgery for patients undergoing vertical sleeve gastrectomy (VSG).
  Apixaban: New Oral Anticoagulants (NOACs) are currently available for prophylaxis against venous thromboembolism in patients undergoing total hip or knee replacement surgery.
Period: Overall Study
Arm/Group | APB Study: Apixaban Pharmacokinetics in RYGB | APB Study: Apixaban Pharmacokinetics in VSG
Started | 17 | 16
Completed | 14 | 14
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APB Study: Apixaban Pharmacokinetics in VSG | APB Study: Apixaban Pharmacokinetics in RYGB | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.6) | 42 (10.2) | 43.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Pharmacokinetics as Assessed by Cmax (Max Concentration)
Description: To determine the durability or change in pharmacokinetics of apixaban in patients with obesity following one of two bariatric surgical procedures. Change in Cmax (ng/ml) between 12 months and baseline.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | APB Study: Apixaban Pharmacokinetics in VSG | APB Study: Apixaban Pharmacokinetics in RYGB
Number analyzed (Participants) | 14 | 14
ng/ml | 5.3 (19.98) | -6.7 (25.35)

2. Primary Outcome: Change in Pharmacokinetics as Assessed by Area Under the Curve (AUC)
Description: To determine the durability or change in pharmacokinetics of apixaban in patients with obesity following one of two bariatric surgical procedures. Change in AUC (ng*h/ml) between 12 months and baseline.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | APB Study: Apixaban Pharmacokinetics in VSG | APB Study: Apixaban Pharmacokinetics in RYGB
Number analyzed (Participants) | 14 | 14
ng*h/ml | -168.25 (226.36) | -166.34 (264.36)

3. Primary Outcome: Change in Pharmacokinetics as Assessed by Elimination Half-life
Description: To determine the durability or change in pharmacokinetics of apixaban in patients with obesity following one of two bariatric surgical procedures.
Time Frame: Baseline and 12 months
Population: This outcome measure was not assessed. Data was not collected.
Arm/Group | APB Study: Apixaban Pharmacokinetics in VSG | APB Study: Apixaban Pharmacokinetics in RYGB
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Pharmacodynamics as Assessed by Factor Xa Levels (Percent Activity)
Description: To determine the durability or change in pharmacodynamics of apixaban in patients with obesity following one of two bariatric surgical procedures. Reported data is the difference between 12 months and baseline. Factor Xa levels is measured in "percent activity".
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Percent Activity
Arm/Group | APB Study: Apixaban Pharmacokinetics in VSG | APB Study: Apixaban Pharmacokinetics in RYGB
Number analyzed (Participants) | 14 | 14
Percent Activity | -7.3 (17.8) | -15.7 (21.03)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | APB Study: Apixaban Pharmacokinetics in RYGB | APB Study: Apixaban Pharmacokinetics in VSG
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/16
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/16
Other Adverse Events (participants affected / at risk) | 1/17 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APB Study: Apixaban Pharmacokinetics in RYGB (N=17) | APB Study: Apixaban Pharmacokinetics in VSG (N=16)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sudden Cardiac Death (Cardiac disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APB Study: Apixaban Pharmacokinetics in RYGB (N=17) | APB Study: Apixaban Pharmacokinetics in VSG (N=16)
migraine headache (General disorders) | 0 (0) | 1 (1)
Zoster Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02406885/Prot_SAP_000.pdf